CLINICAL TRIAL: NCT07271199
Title: Evaluation of the Eyelash Care Effects of Premium Rejuvenation Eyelash Serum
Brief Title: Eyelash Effect Evaluation for Premium Rejuvenation Eyelash Serum
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hungkuang University (Other)
Collaborators: Schweitzer Biotech Company (Unknown)
Responsible Party: Principal Investigator, Tsong-Min Chang, Vice President, Hungkuang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 25-089-A
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Skin Condition; Eyelash Growth; Eyelashes; Skin Health; Hair Health
Keywords: Eyelash; Eyelash health; Skin health; Eyelash condition; Hair health; Product formulation; Growth factors; Extracellular vesicle; Ginger; Turmeric
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Placebo control (Placebo Comparator): Base formula without active ingredient
  Interventions: Other: Placebo control
- Group 2: Experimental formula (Experimental): Base formula with ginger (Zingiber officinale)-derived extracellular vesicle, turmeric (Curcuma longa)-derived extracellular vesicles, insulin growth factor-1 (IGF-1), and fibroblast growth factor-7 (FGF-7).
  Interventions: Other: Experimental formula

INTERVENTIONS:
Other: Placebo control — Placebo Control (Base Formula without active ingredients). After thoroughly cleansing the face and removing contact lenses (if applicable), apply 1 mL of the serum evenly to the base of the eyelashes. Allow the serum to absorb for a few minutes. Repeat application twice daily, in the morning and evening.
  Arms: Group 1: Placebo control
Other: Experimental formula — Base formula with ginger (Zingiber officinale)-derived extracellular vesicle, turmeric (Curcuma longa)-derived extracellular vesicles, insulin growth factor-1 (IGF-1), and fibroblast growth factor-7 (FGF-7).
  After thoroughly cleansing the face and removing contact lenses (if applicable), apply 1 mL of the serum evenly to the base of the eyelashes. Allow the serum to absorb for a few minutes. Repeat this application twice daily, in the morning and evening.
  Arms: Group 2: Experimental formula

SUMMARY:
This study aims to evaluate the efficacy of the Premium Rejuvenation Eyelash Serum on eyelashes and the surrounding periorbital skin. A total of 30 healthy female participants, aged 18 to 60, will be recruited and randomly assigned to two groups receiving different serum formulations. Participants will apply the product twice daily for 112 days (16 weeks), with eyelash and periorbital skin conditions assessed at multiple time points using non-invasive measurements. Key parameters include eyelash density, eyelash length, and overall periorbital skin condition. At the end of the study (Day 112), both participant self-assessments and evaluations by an eyelash specialist will be conducted to assess changes in eyelash and skin condition.

DETAILED DESCRIPTION:
This prospective, randomized, double-blinded, placebo-controlled study aims to investigate the effects of Premium Rejuvenation Eyelash Serum on eyelashes and surrounding periorbital skin. A total of 30 healthy female adults aged 18 to 60 will be enrolled. Inclusion criteria require participants to be free from chronic diseases, major illnesses (including cancer, stroke-related disorders, paralysis, acute myocardial infarction, coronary artery bypass surgery, end-stage renal disease, or major organ/hematopoietic stem cell transplants), and allergic constitutions. Exclusion criteria include current use of medications or eyelash care products.

Participants will be randomly assigned into two groups of 15 each: Group 1 uses placebo (Base formula without active ingredient); Group 2 uses the experimental formula with ginger (Zingiber officinale)-derived extracellular vesicle + turmeric (Curcuma longa)-derived extracellular vesicles + IGF-1 + FGF-7. . Baseline assessments will be conducted prior to product use. Follow-up assessments will occur at Days 28 (4 weeks), 56 (8 weeks), 84 (12 weeks), and 112 (16 weeks). Evaluations will include eyelash density, change in eyelash length, self-reported periorbital skin condition (e.g., swelling, irritation, pigmentation, redness, and allergic reactions), and a questionnaire. Eyelash parameters will be objectively measured using the Canfield Scientific VISIA® Skin Analysis System. At the conclusion of the study (Day 112), both participant self-assessments and evaluations by an eyelash specialist will be conducted to assess eyelash and surrounding skin condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female adults from the age of 18 to 60 years (inclusive).
* Having symptoms of alopecia, baldness, or self-identified with hair thinning.
* Absence of chronic diseases, major illnesses, or allergies.
* Major illnesses include cancer, post-stroke disorders, paralysis, acute myocardial infarction, coronary artery bypass surgery, end-stage renal disease, and major organ transplant or hematopoietic stem cell transplant

Exclusion Criteria:

* Currently taking any medication or using any eyelash care products.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 30 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Eyelash density | Assessment conducted every 28 days from Day 0 to Day 112 (including Day 0 as baseline)
  Assess eyelash density with Canfield VISIA® Skin Analysis system by assigning score from 1 (most dense, thick eyelashes) to 5 (least dense, thin eyelashes). Results will be expressed as percentage of change in eyelash density percentage relative to Day 0.
Eyelash length | Assessment conducted every 28 days from Day 0 to Day 112 (including Day 0 as baseline)
  Assess eyelash length with Canfield VISIA® Skin Analysis system by assigning score from 1 (longest eyelashes) to 5 (shortest eyelashes). Results will be expressed as percentage of change in eyelash length percentage relative to Day 0
Periorbital skin and eye conditional questionnaire | Assessment conducted every 28 days from Day 0 to Day 112 (including Day 0 as baseline)
  Participants will be asked to answer a questionnaire for self-assessment of periorbital skin conditions such as swelling, irritation, pigmentation, redness, and allergic reaction; corneal and retinal conditions including swelling, hyperemia, and allergic reaction will also be self-evaluated.

SECONDARY OUTCOMES:
Participant self-assessment | Day 112 (End of the study period)
  Participants will be asked to fill out an assessment form with score from 0 to 4 for each of the eyelash condition and product feedback evaluated.
Eyelash specialist assessment | Day 112 (End of the study)
  An eyelash specialist will assess and eyelash and periorbital skin condition of the participant and assign a score from 0 to 4 for each of the evaluated items as well as assign a score of Global Aesthetic Improvement Scale (GAIS) from -1 to 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Hungkuang University, Taichung, Taiwan